CLINICAL TRIAL: NCT00573547
Title: A 12-Week Open-Label Trial of Once-Weekly Fluoxetine for the Treatment of Depression in Patients With End-Stage Renal Disease
Brief Title: Open Label Trial of Fluoxetine for the Treatment of Depression in Patients With End Stage Renal Disease
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Principal Investigator decided not to initiate the study.
Sponsor: Creighton University (Other)
Responsible Party: Syed Pirzada Sattar, M.D., Creighton University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-13860
Record Dates: First submitted 2007-12-12; First posted 2007-12-14 (Estimated); Last update posted 2011-08-16 (Estimated); Status verified 2011-08

CONDITIONS: Depression
Keywords: depression; chronic renal failures; end stage renal disease
MeSH Terms: conditions — Depression; Kidney Failure, Chronic | interventions — Fluoxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Fluoxetine — Fluoxetine will be dosed at 90 mg once a week
  Other Names: Prozac

SUMMARY:
The purpose of this study is to test whether once-weekly prozac therapy leads to reduction in depression in patients requiring kidney dialysis.

DETAILED DESCRIPTION:
Once-weekly Prozac is a psychiatric medicine, approved by the FDA for the use in treatment of psychiatric disorders. This study will test whether once-weekly Prozac leads to reduced symptoms of depression. Patients requiring dialysis often report symptoms of depression either due to the presence of major depression, a relatively common psychiatric disorder, or due to depression secondary to kidney failure.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic renal failure and end stage renal disease
* Ongoing need for regular dialysis treatment
* Diagnosis of depression based on DSMIV
* Age tween 19-65 years

Exclusion Criteria:

* Inability to provide informed consent
* Medically or psychiatrically unstable, as defined by requiring inpatient treatment
* Pregnancy, nursing or refusal to use a reliable method of birth control in women
* Patients with known allergy to fluoxetine, or previous treatment failure of fluoxetine

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-02; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Determine the efficacy and tolerability of once-weekly fluoxetine in patients with End Stage Renal Disorder who have been diagnosed with depression | Patients will come in for once weekly visits for 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Syed P Sattar, MD, Principal Investigator — Creighton University Department of Psychiatry
Locations (2):
- United States (2):
  - Creighton Department of Psychiatry, Omaha, Nebraska
  - Creighton University Department of Psychiatry, Omaha, Nebraska